CLINICAL TRIAL: NCT05680792
Title: Evaluation of Pharmacokinetic Interaction Between Nitazoxanide and Atazanavir/Ritonavir in Healthy Volunteers
Brief Title: Pharmacokinetic Interaction Between Nitazoxanide and Atazanavir/Ritonavir in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Principal Investigator, Babatunde Adeagbo, Principal Investigator, Obafemi Awolowo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IPH/OAU/12/1574
Record Dates: First submitted 2022-12-07; First posted 2023-01-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Drug Interaction
Keywords: Nitazoxanide; atazanavir/ritonavir; drug-drug interaction
MeSH Terms: interventions — nitazoxanide; atazanavir, ritonavir drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of nitazoxanide alone (Other): Participants in this arm will receive 1000 mg of nitazoxanide tablets alone
  Interventions: Drug: Nitazoxanide
- Administration of nitazoxanide plus atazanavir/ritonavir (Other): Participants in this arm will receive 1000 mg of nitazoxanide tablets twice daily together with one tablet of atazanavir/ritonavir (300 mg/100 mg) once daily in the morning.
  Interventions: Drug: Nitazoxanide; Drug: Atazanavir/ritonavir

INTERVENTIONS:
Drug: Nitazoxanide — 1000 mg nitazoxanide tablets twice daily. The drug will be administered after meal for 5 days
  Other Names: Netazox
Drug: Atazanavir/ritonavir — 300/100 mg atazanavir/ritonavir tablets in the evening once daily, to be administered after meal for 5 days.
  Arms: Administration of nitazoxanide plus atazanavir/ritonavir

SUMMARY:
The goal of this study is to

1. determine the most effective biological sampling method that best describe the pharmacokinetics nitazoxanide/tizoxanide and to;
2. evaluate the clinical significance of the pharmacokinetics interaction between nitazoxanide (1000mg twice daily) and atazanavir/ritonavir (300mg/100mg).

Participants will be given 1000mg oral nitazoxanide taken twice daily for seven days. After a washout period of three weeks, they will receive 1000mg oral nitazoxanide with atazanavir/ritonavir (taken orally at 300/100 mg). Five millimetres of whole blood or swab or saliva samples will be collected from them at 0.5, 1, 2, 4, 6, 8 and 12 hours after dose on day 1, 5 and 7.

The pharmacokinetic of nitazoxanide when administered alone and alongside atazanavir/ritonavir will be compared to see if concomitant administration of nitazoxanide and atazanavir/ritonavir affect nitazoxanide pharmacokinetics

DETAILED DESCRIPTION:
Nitazoxanide is an antiprotozoal drug with a well-understood and documented safety profile. It was first approved by the US Food and Drug Administration (FDA) in July 2004 for the treatment of diarrhoea caused by Giardia lamblia or Cryptosporidium parvum in adults (≥ 18 years) and paediatrics (1-17 years). Nitazoxanide has also demonstrated in-vitro anti-SARS-CoV-2 activity. A review of in vitro studies reporting the anti-coronavirus activity of nitazoxanide and its active metabolite, tizoxanide, is available. Nitazoxanide was among the three top inhibitors of coronavirus replication, resulting in a reduction of 6 log10 in virus titer with an IC50 of 1.0 µM. The major circulating metabolite of nitazoxanide is tizoxanide, and it has also been confirmed to have activity against SARS-CoV-216. Both suppress the cytopathic effect of SARS-CoV-2. Nitazoxanide is also active against the influenza A virus and was shown to reduce symptom duration in uncomplicated acute influenza. Since SARS-CoV-2 shares almost 80% of the genome with SARSCoV19 and almost all encoded proteins of SARS-CoV-2 are homologous to SARS-CoV proteins, nitazoxanide and its metabolite tizoxanide with demonstrated activity against SARS-CoV are likely to be effective against SARS-CoV-2. Since the virus replicates quickly, antivirals must remain active across their dosing interval. Therefore, enhanced drug concentration will be needed in the lung throughout the dosing interval.

The HIV protease inhibitor, atazanavir (boosted with ritonavir), has been shown to inhibit the major protease enzyme required for viral polyprotein processing during coronavirus replication. It also blocks pro-inflammatory cytokine production. Similar to nitazoxanide, atazanavir has been shown to achieve effective concentration in the pulmonary tissues at the approved dose of 300 mg in combination with 100 mg of ritonavir, with even more favourable ratios when compared to in vitro activities generated in human cell models.

Therefore, based on these considerations, the combination of nitazoxanide (taken orally at 1000 mg twice daily) and atazanavir/ritonavir (taken orally at 300/100 mg once daily) is being considered for selection for intervention for the treatment of COVID-19. Hence, this study wants to evaluate the clinical usefulness of the combination of these drugs. The approach is to characterise the extent of drug-drug interaction of nitazoxanide and atazanavir/ritonavir when 1000 mg nitazoxanide is taken two times daily in combination with 300/100 mg atazanavir/ritonavir before deploying the combination for the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include both male and female healthy volunteers that are eighteen years or above
* non-smokers, non-alcoholics, had not taken any medication or coffee 2 weeks before participating, were non-pregnant and non-breastfeeding

Exclusion Criteria:

* Pregnant women will be excluded from the study. Moreover, volunteers who have been on any other drugs in the last two weeks will also be excluded from the study.
* Exclusion criteria included any sickness or reaction to the study drugs.

Ages: 18 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Minimum plasma concentration (Cmin) | After the first dose (Day 1)
  Tizoxanide minimum plasma concentration with or without atazanavir/ritonavir
Minimum plasma concentration (Cmin) | At Day 5
  Tizoxanide minimum plasma concentration with or without atazanavir/ritonavir
Maximum plasma concentration (Cmax) | After the first dose (Day 1)
  Tizoxanide maximum plasma concentration with or without atazanavir/ritonavir
Maximum plasma concentration (Cmax) | At Day 5
  Tizoxanide maximum plasma concentration with or without atazanavir/ritonavir
Area under the concentration-time curve (AUC) | After the first dose (Day 1)
  Tizoxanide Area under the concentration-time curve with or without atazanavir/ritonavir
Area under the concentration-time curve (AUC) | At Day 5
  Tizoxanide Area under the concentration-time curve with or without atazanavir/ritonavir

CONTACTS AND LOCATIONS:
Overall Officials: Babatunde A Adeagbo, PhD, Principal Investigator — Obafemi Awolowo University
Locations (1):
- Obafemi Awolowo University, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No